CLINICAL TRIAL: NCT03635424
Title: Transcatheter Aortic Valve Replacement (TAVR) With Medtronic TAVR System in Patients With Severe Bicuspid Aortic Valve Stenosis and at Low Predicted Risk of Mortality With Surgical Aortic Valve Replacement (SAVR)
Brief Title: Medtronic Transcatheter Aortic Valve Replacement (TAVR) Low Risk Bicuspid Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10790330DOC
Record Dates: First submitted 2018-07-31; First posted 2018-08-17 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Bicuspid Aortic Valve
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Medtronic TAVR Systems (Experimental): Treatment of patients with bicuspid aortic anatomy and severe aortic stenosis at low risk for SAVR with Medtronic Evolut PRO and Evolut R systems
  Interventions: Device: Medtronic TAVR Systems

INTERVENTIONS:
Device: Medtronic TAVR Systems — Treatment of patients with bicuspid aortic anatomy and severe aortic stenosis at low risk for SAVR with Medtronic Evolut PRO and Evolut R systems

SUMMARY:
The objective of the trial is to evaluate the procedural safety and efficacy of the Medtronic TAVR system in patients with bicuspid aortic anatomy and severe aortic stenosis at low risk for SAVR

DETAILED DESCRIPTION:
Multi-center, prospective, single arm

All subjects will be treated with a Medtronic TAVR system. Subject follow-ups will be conducted at pre and post-procedure, discharge, 30 days, 1 year, and annually through 10 years

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic stenosis, defined as follows:

   1. For symptomatic patients:

      Aortic valve area ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), OR mean gradient ≥40 mmHg, OR Maximal aortic valve velocity ≥4.0 m/sec by transthoracic echocardiography at rest
   2. For asymptomatic patients:

   Very severe aortic stenosis with an aortic valve area of ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), AND maximal aortic velocity ≥5.0 m/sec, or mean gradient ≥60 mmHg by transthoracic echocardiography at rest, OR

   Aortic valve area of ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), AND a mean gradient ≥40 mmHg or maximal aortic valve velocity ≥4.0 m/sec by transthoracic echocardiography at rest, AND an exercise tolerance test that demonstrates a limited exercise capacity, abnormal BP response, or arrhythmia OR

   Aortic valve area of ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), AND mean gradient ≥40 mmHg, or maximal aortic valve velocity ≥4.0 m/sec by transthoracic echocardiography at rest, AND a left ventricular ejection fraction <50%.
2. Patient is considered low risk for SAVR, where low risk is defined as predicted risk of mortality for SAVR <3% at 30 days per multidisciplinary local heart team assessment.
3. Bicuspid aortic valve anatomy (all sub-types) confirmed by MDCT.
4. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

Exclusion Criteria:

1. Any condition considered a contraindication for placement of a bioprosthetic valve (eg, subject is indicated for mechanical prosthetic valve).
2. Age less than 60 years
3. A known hypersensitivity or contraindication to any of the following that cannot be adequately pre-medicated:

   1. aspirin or heparin (HIT/HITTS) and bivalirudin
   2. ticlopidine and clopidogrel
   3. Nitinol (titanium or nickel)
   4. contrast media
4. Blood dyscrasias as defined: leukopenia (WBC <1000 mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states.
5. Ongoing sepsis, including active endocarditis.
6. Any percutaneous coronary or peripheral interventional procedure with a bare metal stent or drug eluting stent performed within 30 days prior to screening committee approval.
7. Multivessel coronary artery disease with a Syntax score >22 and/or unprotected left main coronary artery.
8. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 10 weeks of Heart Team assessment.
9. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
10. Recent (within 2 months of Heart Team assessment) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
11. Gastrointestinal (GI) bleeding that would preclude anticoagulation.
12. Subject refuses a blood transfusion.
13. Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
14. Estimated life expectancy of less than 24 months due to associated non-cardiac co-morbid conditions.
15. Other medical, social, or psychological conditions that in the opinion of the investigator precludes the subject from appropriate consent or adherence to the protocol required follow-up exams.
16. Currently participating in an investigational drug or another device study (excluding registries).
17. Evidence of an acute myocardial infarction ≤30 days before the study procedure due to unstable coronary artery disease (WHO criteria).
18. Need for emergency surgery for any reason.
19. Subject is pregnant or breast feeding.
20. Subject is legally incompetent, or otherwise vulnerable

    Anatomical exclusion criteria:
21. Pre-existing prosthetic heart valve in any position.
22. Severe mitral regurgitation amenable to surgical replacement or repair.
23. Severe tricuspid regurgitation amenable to surgical replacement or repair.
24. Moderate or severe mitral stenosis amenable to surgical replacement or repair.
25. Hypertrophic obstructive cardiomyopathy with left ventricular outflow gradient.
26. Prohibitive left ventricular outflow tract calcification.
27. Sinus of Valsalva diameter unsuitable for placement of the self-expanding bioprosthesis
28. Aortic annulus diameter of <18 or >30 mm.
29. Significant ascending aortopathy requiring surgical repair
30. Ascending aorta diameter > 4.5 cm

    For transfemoral or transaxillary (subclavian) access:
31. Access vessel mean diameter <5.0 mm for Evolut 23R, 26R, or 29R mm TAV, or access vessel mean diameter <5.5 mm for Evolut 34R mm or Evolut PRO 23R, 26R, 29 R mm TAV. However, for transaxillary (subclavian) access in patients with a patent LIMA, access vessel mean diameter <5.5mm for Evolut 23R, 26R, or 29R mm TAV, or access vessel mean diameter <6.0 mm for the Evolut 34R or Evolut PRO TAV.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reardon, MD, Study Chair — The Methodist Hospital Research Institute; John Forrest, MD, Principal Investigator — Yale University; Basel Ramlawi, MD, Principal Investigator — Paramount Heart
Locations (25):
- United States (25):
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - HealthPark Medical Center, Fort Myers, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Spectrum Health Hospital, Grand Rapids, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - North Shore University Hospital, Manhasset, New York
  - The Mount Sinai Hospital, New York, New York
  - Saint Francis Hospital, Roslyn, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - UPMC Pinnacle Harrisburg Campus, Harrisburg, Pennsylvania
  - Paramount Heart, Villanova, Pennsylvania
  - Baylor Jack and Jane Hamilton Heart & Vascular Hospital, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Forrest JK, Ramlawi B, Deeb GM, Zahr F, Song HK, Kleiman NS, Chetcuti SJ, Michelena HI, Mangi AA, Skiles JA, Huang J, Popma JJ, Reardon MJ. Transcatheter Aortic Valve Replacement in Low-risk Patients With Bicuspid Aortic Valve Stenosis. JAMA Cardiol. 2021 Jan 1;6(1):50-57. doi: 10.1001/jamacardio.2020.4738. PMID 33031491

RESULTS

PARTICIPANT FLOW:
Groups:
- Medtronic TAVR Systems: Treatment with Medtronic Evolut PRO and Evolut R systems
Period: Overall Study
Arm/Group | Medtronic TAVR Systems
Started | 150
Completed | 147
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Device not implanted | 1

BASELINE CHARACTERISTICS:
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: Years of age] | 70.3 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  United States | 150
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Calculated surface area of the human body in m^2
  m^2 | 1.9 (0.2)
Society of Thoracic Surgeons (STS) Score [Mean (Standard Deviation); unit: % risk of mortality] — STS score of predicted risk of 30-day mortality
  % risk of mortality | 1.4 (0.6)
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — NYHA Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Participants
    NYHA Class I | 3
    NYHA Class II | 106
    NYHA Class III | 40
    NYHA Class IV | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety: Percent of Participants With All-Cause Mortality or Disabling Stroke Rate at 30 Days Post-procedure.
Description: Rate of of all-cause mortality or disabling stroke rate at 30 days
Time Frame: 30 days
Population: Attempted Implant Set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Percent of participants (K-M rate) | 1.3

2. Primary Outcome: Efficacy: Percent of Participants Who Meet All Device Success Criteria at 30 Days Post-procedure.
Description: Device success rate, defined as:
  * Absence of procedural mortality, AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location, AND
  * Absence of moderate or severe total prosthetic valve regurgitation (at 18 hours to 7 days)
Time Frame: 7 days
Population: Implanted Set
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 148
Percent of participants | 95.9 [91.3 to 98.5]

3. Secondary Outcome: All-Cause Mortality Rate
Description: Rate of all cause mortality
Time Frame: 1 year and annually through 10 years
Reporting Status: Not Posted

4. Secondary Outcome: All Stroke (Disabling and Non-Disabling) Rate
Description: Rate of disabling and non-disabling strokes
Time Frame: 1 year and annually through 10 years
Reporting Status: Not Posted

5. Secondary Outcome: Percent of Participants With New Permanent Pacemaker Implantation at 30 Days Post-procedure.
Description: Rate of new permanent pacemaker implantation at 30 days post-procedure (excludes patients with pre-existing pacemaker at baseline)
Time Frame: 30 days
Population: Attempted Implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Percent of participants (K-M rate) | 15.1

6. Secondary Outcome: Percent of Participants Who Experience a Myocardial Infarction at 30 Days Post-procedure.
Description: The rate of myocardial infarction at 30 days
Time Frame: 30 days
Population: Attempted Implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Percent of participants (K-M rate)
  Myocardial infarction | 0.7
  Peri-procedural myocarial infarction | 0.0
  Spontaneous myocardial infarction | 0.7

7. Secondary Outcome: Percent of Participants With a Life-Threatening Bleeding Event at 30 Days Post-procedure.
Description: Rate of life-threatening (or disabling) bleeding at 30 days
Time Frame: 30 days
Population: Attempted Implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Percent of participants (K-M rate) | 4.0

8. Secondary Outcome: Percent of Participants With Prosthetic Valve Endocarditis at 30 Days Post-procedure.
Description: Rate of prosthetic valve endocarditis at 30 days
Time Frame: 30 days
Population: Attempted Implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Percent of participants (K-M rate) | 0.0

9. Secondary Outcome: Percent of Participant With Prosthetic Valve Thrombosis at 30 Days Post-procedure.
Description: Rate of prosthetic valve thrombosis at 30 days
Time Frame: 30 days
Population: Attempted Implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Percent of participants (K-M rate) | 0.7

10. Secondary Outcome: Percent pf Participants With Valve-Related Dysfunction Requiring Repeat Procedure at 30 Days Post-procedure.
Description: Rate of valve-related dysfunction requiring repeat procedure at 30 days
Time Frame: 30 days
Population: Attempted Implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Percent of participants (K-M rate) | 0.0

11. Secondary Outcome: Percent of Participants With a Repeat Hospitalization for Aortic Valve Disease at 30 Days Post-procedure.
Description: Rate of repeat hospitalization for aortic valve disease at 30 days
Time Frame: 30 days
Population: Attempted Implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Percent of participants (K-M rate) | 4.0

12. Secondary Outcome: Percent of Participants With a Repeat Hospitalization for Ascending Aorta Disease at 30 Days Post-procedure.
Description: Rate of repeat hospitalization for ascending aorta disease at 30 days
Time Frame: 30 days
Population: Attempted Implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Percent of participants (K-M rate) | 0.0

13. Secondary Outcome: Hemodynamic Performance Metrics by Doppler Echocardiography: Mean Aortic Gradient Reported as Mean Average at Baseline and 30 Days
Description: Reporting of prosthetic valve hemodynamic performance by transvalvular mean aortic gradient
Time Frame: 30 days
Population: Implanted set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 148
mmHg
  Baseline | 48.01 (16.09)
  30 Day | 7.58 (3.69)

14. Secondary Outcome: Hemodynamic Performance Metrics by Doppler Echocardiography: Effective Orifice Area Reported as Mean Average at Baseline and 30 Days.
Description: Change in hemodynamic performance metrics by Doppler echocardiography measured by effective orifice area.
Time Frame: 30 days
Population: Implanted set
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 148
cm^2
  Baseline | 0.81 (0.23)
  30 Day | 2.28 (0.73)

15. Secondary Outcome: Hemodynamic Performance Metrics by Doppler Echocardiography: Percent of Participants With Degrees of Total Prosthetic Valve Regurgitation at Baseline and 30 Days
Description: Reporting of prosthetic valve hemodynamic performance by degree of total prosthetic valve regurgitation at 30 days post-procedure
Time Frame: 30 days
Population: Implanted set
Measure: Number; unit: Percentage of participants
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 148
Percentage of participants
  Baseline: None | 30.4
  Baseline: Trace | 24.3
  Baseline: Mild/Mild to Moderate | 42.6
  Baseline: Moderate/Moderate to Severe | 2.7
  Baseline: Severe | 0.0
  Baseline: >=Moderate | 2.7
  30 Day: None | 34.2
  30 Day: Trace | 25.3
  30 Day: Mild/Mild to Moderate | 40.4
  30 Day: Moderate/Moderate to Severe | 0.0
  30 Day: Severe | 0.0
  30 Day: >=Moderate | 0.0

16. Secondary Outcome: Hemodynamic Performance Metrics by Doppler Echocardiography: Percent of Participants With Degrees of Paravalvular Prosthetic Regurgitation at 30 Days
Description: Reporting of prosthetic valve hemodynamic performance by degree of paravalvular regurgitation at 30 days post-procedure
Time Frame: 30 days
Population: Implanted set
Measure: Number; unit: Percentage of participants
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 148
Percentage of participants
  30 Day: None | 36.1
  30 Day: Trace | 23.6
  30 Day: Mild/Mild to Moderate | 40.3
  30 Day: Moderate/Moderate to Severe | 0.0
  30 Day: Severe | 0.0
  30 Day: >=Moderate | 0.0

17. Secondary Outcome: Hemodynamic Performance Metrics by Doppler Echocardiography: Percent of Participants With Degrees of Transvalvular Prosthetic Regurgitation at 30 Days
Description: Reporting of prosthetic valve hemodynamic performance by degree of transvalvular regurgitation at 30 days post-procedure
Time Frame: 30 days
Population: Implanted set
Measure: Number; unit: Percentage of participants
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 148
Percentage of participants
  30 Day: None | 95.1
  30 Day: Trace | 4.9
  30 Day: Mild/Mild to Moderate | 0.0
  30 Day: Moderate/Moderate to Severe | 0.0
  30 Day: Severe | 0.0
  30 Day: >=Moderate | 0.0

18. Secondary Outcome: New York Heart Association (NYHA) Functional Classification at Baseline and 30 Days
Description: Reporting of NYHA classification change from baseline to 30 days
  NYHA Classification criteria:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
Time Frame: 30 days
Population: Attempted Implant set
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 147
Participants
  30 day - Improved | 121
  30 day - No Change | 23
  30 day - Worsened | 2
  30 day - Died | 1

19. Secondary Outcome: Change in Health-related Quality of Life (QoL) as Assessed by Kansas City Cardiomyopathy (KCCQ) Instrument at Baseline and 30 Days
Description: QoL overall summary (all domains below) and clinical summary (physical function and symptoms only) scores and change in summary scores from baseline using the following measures:
  • KCCQ: Quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: 30 days
Population: Attempted Implant set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Score on a scale
  Baseline KCCQ - Overall | 68.5 (19.6)
  Baseline KCCQ - Clinical | 73.7 (20.3)
  30 day KCCQ - Overall | 90.3 (12.8)
  30 day KCCQ - Clinical | 91.3 (12.5)
  30 day change from baseline KCCQ - Overall | 21.6 (17.6)
  30 day change from baseline KCCQ - Clinical | 17.6 (17.7)

20. Secondary Outcome: Health-related Quality of Life (QoL) as Assessed by European QoL (EQ-5D) at Baseline and 30 Days.
Description: QoL summary scores and change from baseline using the following measures:
  • EQ-5D: Measures 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that can be converted to utilities using an algorithm. Utilities range from 0 to 1, with 1 representing perfect health, and 0 corresponding to the worst imaginable health state
Time Frame: 30 days
Population: Attempted Implant set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Medtronic TAVR Systems
Number analyzed (Participants) | 150
Score on a scale
  Baseline EQ-5D Index Score | 0.8 (0.1)
  30 day EQ-5D Index Score | 0.9 (0.1)
  30 day change from baseline EQ-5D Index Score | 0.1 (0.1)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from study enrollment through the 2 year follow-up visit. Adverse event data are currently available and reported for up to 30 days post-procedure.
Description: All new or worsening AEs will be collected through 2 years. After 2 years only serious and device-related events will be collected.
Arm/Group | Medtronic TAVR Systems
All-Cause Mortality (participants affected / at risk) | 1/150
Serious Adverse Events (participants affected / at risk) | 57/150
Other Adverse Events (participants affected / at risk) | 120/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic TAVR Systems (N=150)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Atrial Flutter (Cardiac disorders) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 2 (2)
Atrioventricular Block Complete (Cardiac disorders) | 13 (13)
Atrioventricular Block Second Degree (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2)
Bundle Branch Block Left (Cardiac disorders) | 5 (5)
Bundle Branch Block Right (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Conduction Disorder (Cardiac disorders) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Hemangioma Congenital (Congenital, familial and genetic disorders) | 1 (1)
Retinal Artery Occlusion (Eye disorders) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2 (2)
Chest Discomfort (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Device Embolization (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pneumonia Klebsiella (Infections and infestations) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Device Deployment Issue (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Site Complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Embolic Stroke (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Device Leakage (Product Issues) | 4 (4)
Device Malfunction (Product Issues) | 1 (1)
Acute Pulmonary Edema (Reproductive system and breast disorders) | 1 (1)
Acute Respiratory Failure (Reproductive system and breast disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Femoral Artery Dissection (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 7 (7)
Peripheral Artery Stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic TAVR Systems (N=150)
Anemia (Blood and lymphatic system disorders) | 10 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (13)
Atrioventricular Block First Degree (Cardiac disorders) | 18 (19)
Bundle Branch Block Left (Cardiac disorders) | 51 (51)
Bundle Branch Block Right (Cardiac disorders) | 9 (9)
Anemia Postoperative (Injury, poisoning and procedural complications) | 8 (8)
Hypertension (Vascular disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 60 days of receipt Medtronic (MDT) will verify presence of Confidential Information (CI) & won't censor or interfere with presentation/conclusions except to protect CI (other than Study Data) & its rights in patentable or copyrightable materials, & check technical accuracy of MDT data. If told by MDT that Publication contains CI or technical errors of MDT data, PI will make requested changes before publishing/presenting. PI will delay publication up to 90 more days, if requested.

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/24/NCT03635424/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT03635424/SAP_001.pdf